CLINICAL TRIAL: NCT03317626
Title: Gravity Flow Technique to Validate Proper Location of Epidural Needle Tip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-00975
Record Dates: First submitted 2017-10-17; First posted 2017-10-23 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Epidural Anesthesia
MeSH Terms: interventions — Ice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cold Stimulus (Experimental): The study procedure will beto use a coldstimulus (ice) to assess the subjects for hypesthesia the dermatomes of the lower abdomen at 15 minutes and if necessary at 30 minutes after the epidural is inserted
  Interventions: Diagnostic Test: Cold Stimulus (ice) Test

INTERVENTIONS:
Diagnostic Test: Cold Stimulus (ice) Test — Standard of care epidural will be inserted. The study procedure will be to use a cold stimulus (ice) to assess the subjects for hypesthesia the dermatomes of the lower abdomen at 15 minutes and if necessary at 30 minutes after the epidural is inserted. Hypesthesia to cold will be taken a sign of successful lumbar epidural block.

SUMMARY:
Epidural analgesia for childbirth may fail to provide adequate pain relief. At NYULMC, to maximize the likelihood that epidural analgesia will work well, the gravity flow technique is used when performing epidural procedures.

The gravity flow technique is not well known, and is therefore used in only a few hospitals. The purpose of this study is to quantify the reliability of the gravity flow technique to accurately validate the position of the epidural needle tip when performing lumbar epidural analgesia in laboring women.

DETAILED DESCRIPTION:
The purpose of this study is to quantify the reliability of the gravity flow technique to accurately validate the position of the epidural needle tip when performing lumbar epidural analgesia in laboring women. This gravity flow technique was first described 26 years ago in 1991, and has been at NYU Langone for 15 years, since 2002. The technique has not been formally studied and this study is designed to enable assessment of the success rate of the gravity flow technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients requesting epidural analgesia for labor
* ASA physical status I to II
* Ability to speak and read English to fully comprehend the consent process

Exclusion Criteria:

* Combined spinal-epidural anesthesia
* Coagulopathy
* History of lumbar spine surgery
* Allergy or contraindication to any of the study medications
* Contraindication to epidural analgesia
* ASA physical status >III

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women who have requested epidural analgesia for childbirth
Enrollment: 100 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2018-02-05 (Actual)

PRIMARY OUTCOMES:
Accurate validation of the position of the epidural needle tip whenperforming lumbar epidural analgesia in laboring women. | 30 Minutes post intervention
  Success will be defined as a bilateral decrease of sensation (hypesthesia) to cold and ice in at least 2 adjacent dermatomes between T8 and L2

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Grant, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States